CLINICAL TRIAL: NCT06202365
Title: Acute Effect of Whole Body Vibration on Trunk Endurance and Balance in Obese Female Students
Brief Title: Whole Body Vibration in Obese Female Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Approval No. 2023-125
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Obesity
Keywords: Whole body vibration; Trunk endurance; Balance; Obesity; Females
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (WBV Group) (Experimental): A vibrating platform (WBV) will be used in this study with 6 training exercises for 4 minutes, 2 times /week for 6 weeks. Feet should be parallel at shoulder width apart and knees hold constant. WBV sessions were conducted from low to medium-vibration mode
  Interventions: Device: Whole body Vibration
- Group B (Sham WBV Group) (Sham Comparator): They will receive the same intervention while the device turned off for 4 minutes, 2 session/ week for 6 weeks.
  Interventions: Other: Sham Whole body vibration

INTERVENTIONS:
Device: Whole body Vibration — A vibrating platform (WBV) will be used in this study with 6 training exercises for 4 minutes, 2 times /week for 6 weeks. Feet should be parallel at shoulder width apart and knees hold constant. WBV sessions were conducted from low to medium-vibration mode
  Arms: Group A (WBV Group)
Other: Sham Whole body vibration — They will receive the same intervention while the device turned off for 4 minutes, 2 times /week for 6 weeks.
  Arms: Group B (Sham WBV Group)

SUMMARY:
Obesity is a global public-health issue, with rising incidence and prevalence, significant expenditures, and poor results. Obesity has become a worldwide epidemic in both developed and underdeveloped countries. A body mass index (BMI) of 30 kg/m2 is required for class I obesity, a BMI of 35 - 39.9 kg/m2 is required for class II obesity, and a BMI of 40 kg/m2 is required for class III obesity (morbidly obese). Obesity will be the likely situation for the majority of the adult population during the next two decades due to an abundance of calorie-rich food and apathy toward exercise.

DETAILED DESCRIPTION:
Obese and overweight young people swayed at a higher rate than people of normal weight. Two hypotheses have been offered to explain the negative effect of weight on balance control. The first is decreased plantar sensitivity as a result of hyper-activation of plantar mechanoreceptors caused by the constant pressure of supporting a heavy burden. The second theory is that there is a higher mechanical demand owing to the big body mass itself, as well as a non-negligible amount of body mass further away from the axis of rotation (i.e., ankle joint in an inverted pendulum model) that creates a higher gravitational torque. As a result, in order to maintain an upright posture, the gravitational torque that accelerates the body must be opposed by muscle torques.

WBV is a mechanical stimulation characterized by oscillatory motion supplied from a platform to the entire body. The current devices employ two distinct systems: (a) a vertical vibration, in which the entire plate oscillates uniformly up and down with only a vertical translation; and (b) reciprocating vertical displacements on the left and right sides of a fulcrum, which increases the lateral accelerations. WBV training includes biomechanical characteristics such as body position, amplitude, frequency, magnitude, and duration.

ELIGIBILITY:
Inclusion Criteria:

* Female students
* BMI ≥ 30
* Aged from 18 to 25 years old

Exclusion Criteria:

* Pregnancy
* Musculoskeletal disorders
* History of spinal surgery
* Epilepsy
* Medications that could affect the musculoskeletal system
* Performing regular exercise of more than 3 times a week
* Metal plates in the body
* Ligament sprain
* Medical history such as cardiovascular disease, or diabetes mellitus

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female Students
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Sorensen Test | 6 weeks
  The participants will be asked to lie prone on the treatment table with their hips and knees extended and their arms crossed over their chest, then placing a strap over the pelvis, knees and ankles for support. Then they will be instructed to raise their upper body off the table until their back were parallel to the floor

SECONDARY OUTCOMES:
Trunk flexor endurance Test | 6 weeks
  The participants will be asked to maintain supine position on the examination table. The lower extremities will be positioned comfortably with the knees flexed, and the feet up. The arms will be placed over the chest or behind the head 6 without pulling on the neck. They will be instructed to perform a partial or full sit-up, engaging the trunk flexors to lift the upper body off the surface.
Single leg test | 6 weeks
  for assessment of static balance, the participants will be asked to stand on the dominant leg with their arms crossed over the chest and closed eyes. Then the time will be counted while maintaining this position.
Dynamic balance | 6 weeks
  the Biodex Balance System (BBS) SD (12.1-inch [30.7-cm] display, 115 VAC; Biodex Medical Systems Inc., Shirley, NY, USA). The BBS measures stability indices, which represent the variance of foot platform displacement in degrees for motion in different planes. The platform is fixable and movable.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M Eladl, PhD, Study Director — Assisstant professor of physical therapy for surgery, Faculty of physical therapy
Locations (1):
- Nesma Morgan Allam, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No